CLINICAL TRIAL: NCT00770666
Title: Flexibly-Dosed Combination Pharmacotherapy Versus Standard-Dosed Nicotine Patch Alone for Smokers With Medical Illness
Brief Title: Combination Medications vs. Patch Alone for Medically-Ill Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Michael Steinberg, MD, MPH, UMDNJ-Robert Wood Johnson Medical School
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0220055373
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-10

CONDITIONS: Smoking Cessation
Keywords: Tobacco dependence treatment
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nicotine patch, nicotine inhaler, bupropion
  Interventions: Drug: Nicotine patch, nicotine inhaler, bupropion
- 2 (Active Comparator): Nicotine patch
  Interventions: Drug: Nicotine patch

INTERVENTIONS:
Drug: Nicotine patch, nicotine inhaler, bupropion — Patch - 21 mg - taper as able Inhaler - as needed Bupropion SR 150 mg daily
  Arms: 1
Drug: Nicotine patch — 21 mg daily for 6 weeks followed by 14 mg for 2 weeks and then 7 mg for 2 weeks
  Arms: 2

SUMMARY:
Randomized clinical trial to evaluate a flexibly-dosed-3-medication combination for up to 6 months in smokers with medical illness

DETAILED DESCRIPTION:
Subjects randomly received either nicotine patch alone for a 10-week, tapering course (n=64) or the combination of nicotine patch, nicotine oral inhaler, and bupropion for an ad-lib duration (n=63).

ELIGIBILITY:
Inclusion Criteria:

* currently smoking at least 10 cigarettes per day (confirmed by high exhaled carbon-monoxide (CO))
* 18 years or older
* interested in quitting within the next 30 days
* one or more pre-defined medical illnesses (including cardiovascular disease, other vascular disease, chronic pulmonary disease, cancer, hypertension, diabetes, hyperlipidemia, and recurrent pulmonary infections)

Exclusion Criteria:

* contraindications to pharmacotherapy (including unstable angina, myocardial infarction within 2 months, severe arrhythmia, seizure disorder, serious mental illness requiring antipsychotic medications)
* current use of other tobacco products (smokeless tobacco, cigars, pipes, etc.), bupropion, clonidine, nortriptyline, or nicotine replacement medications
* unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Tobacco use abstinence | 26 week

SECONDARY OUTCOMES:
Time to first relapse | varies
Duration of medication use | 26 weeks
Adverse clinical events | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Steinberg, MD, MPH, Principal Investigator — UMDNJ-RWJMS
Locations (1):
- Umdnj-Rwjms, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Steinberg MB, Greenhaus S, Schmelzer AC, Bover MT, Foulds J, Hoover DR, Carson JL. Triple-combination pharmacotherapy for medically ill smokers: a randomized trial. Ann Intern Med. 2009 Apr 7;150(7):447-54. doi: 10.7326/0003-4819-150-7-200904070-00004. PMID 19349630